CLINICAL TRIAL: NCT02447978
Title: Duration of Protection Following Five Doses of GlaxoSmithKline's (GSK's) DTaP Vaccines in School Age Children
Brief Title: Duration of Protection: GSK DTaP Vaccines
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201477
Record Dates: First submitted 2015-03-26; First posted 2015-05-19 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Diphtheria; Acellular Pertussis; Tetanus
MeSH Terms: conditions — Diphtheria; Tetanus | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines; PEDIARIX; DTPP vaccine

GROUPS / COHORTS (3):
- PCR-positive pertussis cases: Cases will be all individuals who tested PCR-positive for pertussis and negative for parapertussis during the study period and who received 5 doses of DTaP vaccines (either manufactured by GSK or any brand, depending on study objective) through 84 months of age before testing PCR-positive.
  Interventions: Biological: Infanrix; Biological: Pediarix; Biological: Kinrix
- PCR-negative pertussis controls: Controls will consist of persons who tested PCR-negative for both pertussis and parapertussis and who received 5 DTaP doses (either manufactured by GSK or any brand, depending on study objective) before testing PCR negative.
  Interventions: Biological: Infanrix; Biological: Pediarix; Biological: Kinrix
- KPNC-matched controls: Controls will consist of all KPNC members of the same sex, age (year and quarter of birth), race or ethnic group (7 groups; 6 for reported, 1 for imputed), and medical centre as each pertussis case and who were members on the date the case tested PCR-positive (anchor date).
  Interventions: Biological: Infanrix; Biological: Pediarix; Biological: Kinrix

INTERVENTIONS:
Biological: Infanrix — Diphtheria and Tetanus Toxoids and Acellular Pertussis Vaccine Adsorbed Indicated as a 5-dose series in infants and children 6 weeks to 7 years of age.
Biological: Pediarix — Diphtheria and Tetanus Toxoids and Acellular Pertussis Ad-sorbed, Hepatitis B (Recombinant) and Inactivated Poliovirus Vaccine Indicated as a 3-dose series in infants born of hepatitis B surface antigen (HBsAg)-negative mothers. PEDIARIX may be given as early as 6 weeks of age through 6 years of age (prior to the 7th birthday).
Biological: Kinrix — Diphtheria and Tetanus Toxoids and Acellular Pertussis Ad-sorbed and Inactivated Poliovirus Vaccine

SUMMARY:
The purpose of this study is to assess duration of protection for GSK DTaP vaccines in preventing pertussis.

ELIGIBILITY:
Inclusion Criteria:

* Kaiser Permanente Northern California (KPNC) member who received 5 doses of acellular pertussis vaccines be-tween ages 1 month and 84 months at KPNC.
* The 5th dose was given between the ages of 47 and 84 months.
* All 5 DTaP doses received were manufactured by GSK, depending on study objective (otherwise this criterion will not apply).
* Born in 1999 and later.

Inclusion criteria for cases:

• All individuals meeting above inclusion criteria who tested PCR-positive for pertussis and negative for parapertussis during the study period.

Inclusion criteria for PCR-negative controls:

• All individuals meeting above inclusion criteria who tested PCR-negative for both pertussis and parapertussis during the study period.

Inclusion criteria for KPNC-matched controls:

* All individuals from the general KPNC population meeting above inclusion criteria who match a PCR-positive case on sex, age, race or ethnic group, and medical center.
* KPNC members on the day their matched case under-went the PCR test (anchor date).

Exclusion Criteria:

* Individuals whose PCR test date (or anchor date) is less than 2 weeks after receiving their 5th DTaP dose.
* Individuals who were not KPNC members for greater than 3 months between their 5th DTaP dose and PCR test date (or anchor date).
* Individuals who received reduced antigen content pertussis vaccine (Tdap) or any pertussis-containing vaccine after their 5th DTaP dose but before their PCR test date (or anchor date).

Exclusion criteria for controls:

• Individuals will be excluded from serving as a control once they test positive for pertussis.

Ages: 47 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Kaiser Permanente Northern California (KPNC) member who received 5 doses of acellular pertussis vaccines between ages 1 month and 84 months at KPNC.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Estimated GSK-only DTaP relative decrease in protection against pertussis disease (PCR-confirmed) | Between 1 and 84 months of age of the subjects who received all 5 doses of DTaP (GSK-only) vaccine
  Estimation done by comparing time since the 5th DTaP dose between PCR-positive cases and PCR-negative controls
Estimated DTaP (any brand) relative decrease in protection against pertussis disease (PCR-confirmed) | Between 1 and 84 months of age of the subjects who received all 5 doses of DTaP (any brand) vaccine
  Estimation done by comparing time since the 5th DTaP dose between PCR-positive cases and PCR-negative controls

SECONDARY OUTCOMES:
Estimated GSK-only DTaP relative decrease in protection against pertussis disease (PCR-confirmed) | Between 1 and 84 months of age of the subjects who received all 5 doses of DTaP (GSK-only) vaccine
  Estimation derived from comparing PCR-positive cases and matched controls
Estimated DTaP (any brand) relative decrease in protection against pertussis disease (PCR-confirmed) | Between 1 and 84 months of age of the subjects who received all 5 doses of DTaP (any brand) vaccine
  Estimation derived from comparing PCR-positive cases and matched controls

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Klein NP, Bartlett J, Fireman B, Aukes L, Buck PO, Krishnarajah G, Baxter R. Waning protection following 5 doses of a 3-component diphtheria, tetanus, and acellular pertussis vaccine. Vaccine. 2017 Jun 8;35(26):3395-3400. doi: 10.1016/j.vaccine.2017.05.008. Epub 2017 May 12. PMID 28506516